CLINICAL TRIAL: NCT01034540
Title: A Double-blind, Randomized, Placebo-controlled, Crossover Trial to Assess the Effects of 4 g/d Prescription Omega-3 Acid Ethyl Esters on Indices of Glucose Homeostasis and Lipoprotein Lipids in Subjects With Hypertriglyceridemia
Brief Title: Effects of Prescription Omega-3 Acids on Glucose and Lipoprotein Lipids in Subjects With Hypertriglyceridemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Provident Clinical Research (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Kevin C. Maki, PhD, Study Director/Chief Science Officer, Provident Clinical Research
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PRV-09009
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Results first posted 2013-10-22 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- POM3 (Experimental): POM3 for the first six weeks of treatment. Placebo for the second six weeks of treatment
  Interventions: Drug: POM3
- Placebo (Placebo Comparator): Placebo for the first six weeks of treatment. POM3 for the second six weeks of treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: POM3 — 4 g/day
  Other Names: Lovaza; prescription omega-3 acid ethyl esters
  Arms: POM3
Drug: Placebo — matching placebo capsule, 4 g/day
  Arms: Placebo

SUMMARY:
The objectives of this study are to assess the effects of 4 g/d prescription omega-3 acid ethyl esters (POM3), compared with a placebo, on indices of insulin sensitivity and secretion, as well as aspects of the fasting and postprandial lipid and lipoprotein profiles, in subjects with hypertriglyceridemia.

DETAILED DESCRIPTION:
This trial will utilize a randomized, double-blind, two-period crossover design. At Visit 2 (Week 0), subjects meeting all entry criteria will be randomized to one of two treatment sequences: placebo or POM3 for the first 6 week phase followed by the study product they did not receive during the first phase (POM3 or placebo) for the second 6 weeks. There will be a 2-week washout period between treatment phases.

ELIGIBILITY:
Inclusion Criteria:

* Men and postmenopausal women, ages 18-79 years.
* Fasting, triglyceride (TG) level in the borderline high to high range.
* Fasting, low density lipoprotein cholesterol (LDL-C) below the very high range while on no lipid altering therapy or while taking stable-dose statin therapy
* Provide written informed consent and authorization for protected health information

Exclusion Criteria:

* Use of any lipid-altering medications, which cannot be stopped, except stable dose statin therapy.
* Use of any omega-3 fatty acid ethyl ester medications or dietary supplements with >1.0 g/d of eicosapentaenoic acid (EPA), docosahexaenoic acid (DHA), or a combination of EPA and DHA
* coronary heart disease (CHD) or a CHD risk equivalent
* Body mass index over 45 kg per square meter
* Allergy or sensitivity to omega-3 fatty acids, corn or corn products (e.g., corn oil), D-alpha tocopherol (vitamin E) or any ingredients in the study drug
* Certain muscle, liver, kidney, lung or gastrointestinal conditions
* Poorly controlled hypertension
* Certain medications
* Active cancers treated within prior 2 years (except non-melanoma skin cancer)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C. Maki, PhD, Study Director — Provident Clinical Research
Locations (1):
- Provident Clinical Research (now Biofortis), Addison, Illinois, United States

REFERENCES:
- [Result] Maki KC, Lawless AL, Kelley KM, Dicklin MR, Schild AL, Rains TM. Prescription omega-3-acid ethyl esters reduce fasting and postprandial triglycerides and modestly reduce pancreatic beta-cell response in subjects with primary hypertriglyceridemia. Prostaglandins Leukot Essent Fatty Acids. 2011 Sep-Oct;85(3-4):143-8. doi: 10.1016/j.plefa.2011.06.005. Epub 2011 Jul 19. PMID 21775113

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted using the research clinic database and print advertisements. First subject screened in May 2010 and screening ended in August 2010.
Groups:
- Prescription Omega-3 Acid Ethyl Esters/Placebo: Prescription omega-3 acid ethyl esters (POM3; Lovaza 4 g/d) for the first six weeks of treatment. Placebo (corn oil 4 g/d) for the second six weeks of treatment
- Placebo/Prescription Omega-3 Acid Ethyl Esters: Placebo (corn oil 4 g/d) for the first six weeks of treatment. Prescription omega-3 acid ethyl esters (POM3; Lovaza 4 g/d) for the second six weeks of treatment
Period: Overall Study
Arm/Group | Prescription Omega-3 Acid Ethyl Esters/Placebo | Placebo/Prescription Omega-3 Acid Ethyl Esters
Started | 11 | 12
Completed 1st Treatment Intervention | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline/adverse event analyses reported for safety population (all randomized subjects who consumed at least 1 dose of study product; n=23). Outcome measures reported for per protocol population (excluded subjects with poor compliance, protocol violations, or without at least 1 outcome data point during each treatment intervention n=19).
Groups:
- Prescription Omega-3 Acid Ethyl Esters (POM3)/Placebo: POM3 for the first six weeks of treatment. Placebo for the second six weeks of treatment
- Placebo/Prescription Omega-3 Acid Ethyl Esters (POM3): Placebo for the first six weeks of treatment. POM3 for the second six weeks of treatment
- Total: Total of all reporting groups
Arm/Group | Prescription Omega-3 Acid Ethyl Esters (POM3)/Placebo | Placebo/Prescription Omega-3 Acid Ethyl Esters (POM3) | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (5.0) | 60.0 (1.7) | 54.2 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Treatments in Liquid Meal Tolerance Test (LMTT) Matsuda Insulin Sensitivity Index (MISI).
Description: Liquid meal tolerance test (LMTT) = two 8 oz servings of Ensure (Abbott Nutrition) + study product followed by blood sample collection at -5, -1, 30, 60, 90, 120, 180, and 240 min, where t = 0 was start of liquid meal consumption. MISI calculated as 10,000/square root of (pre-meal glucose x pre-meal insulin x mean 120 min post-meal glucose x mean 120 min post-meal insulin)
Time Frame: End of Treatment Intervention Period I (week 6) and End of Treatment Intervention Period II (week 14)
Population: Per protocol population in which subjects with poor compliance, protocol violations, and without at least one post-randomization outcome data point during each treatment intervention period were removed.
Measure: Median (Inter-Quartile Range); unit: Index value
Groups:
- Control; Prescription Omega-3 Acid Ethyl Esters: Data from the two treatment sequences (Control/Prescription omega-3-acid ethyl esters and Prescription omega-3-acid ethyl esters/Control) were pooled. Data for treatment intervention period I were collected at week 6; data for treatment intervention period II were collected at week 14.
Arm/Group | Control | Prescription Omega-3 Acid Ethyl Esters
Number analyzed (Participants) | 19 | 19
Index value | 3.2 [1.9 to 7.1] | 3.3 [2.0 to 7.4]
Statistical Analysis 1: Comparison: Control vs Prescription Omega-3 Acid Ethyl Esters; An evaluable sample of 19 subjects provided 80% power (5% alpha-level, 2-tailed) to detect a 2.1 unit difference between control and active in MISI, assuming a 3.0 unit standard deviation (SD). Repeated measures ANOVA was used to assess responses to treatment. Initial repeated measures models contained terms of treatment period, and sequence as fixed effects, with subject modeled as random effect; models were reduced until only significant terms or treatment remained; Test type: Superiority or Other; p = 0.959, ANOVA — Values were not normally distributed, thus analyses were performed on ranked values and medians (IQL) are presented; All tests of statistical significance were completed at the 5% level, two-tailed (p<0.05)

2. Secondary Outcome: Difference Between Treatments in LMTT Insulin Secretion Index and Disposition Index.
Description: Insulin secretion index = total area under the curve from 0 to 120 min post-meal for plasma insulin divided by total area under the curve from 0 to 120 min post-meal for plasma glucose.
  Disposition index = MISI x insulin secretion index
Time Frame: End of Treatment Intervention Period I (week 6) and End of Treatment Intervention Period II (week 14)
Population: Per protocol population excluding subjects with poor compliance and protocol violations.
Measure: Mean (Standard Error); unit: Index value
Groups:
- Control; Prescription Omega-3 Acid Ethyl Esters: Data from the two treatment sequences (Control/Prescription omega-3-acid ethyl esters and Prescription omega-3-acid ethyl esters/Control) were pooled. Treatment period I was the average of values at weeks 4 and 6; treatment period II was the average of values at weeks 12 and 14.
Arm/Group | Control | Prescription Omega-3 Acid Ethyl Esters
Number analyzed (Participants) | 19 | 19
Index value
  Disposition index | 2.4 (0.25) | 2.1 (0.20)
  Insulin secretion index | 0.73 (0.09) | 0.66 (0.09)
Statistical Analysis 1: Comparison: Control vs Prescription Omega-3 Acid Ethyl Esters; Test type: Superiority or Other; p = 0.037, ANOVA; All tests of statistical significance were completed at the 5% level, two-tailed (p<0.05)
Statistical Analysis 2: Comparison: Control vs Prescription Omega-3 Acid Ethyl Esters; Test type: Superiority or Other; p = 0.073, ANOVA — All tests of statistical significance were completed at the 5% level, two-tailed (p<0.05)

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: Adverse event analyses reported for safety population (all randomized subjects who consumed at least 1 dose of study product)
Groups:
- POM3; Placebo: Data from the 2 treatment sequences (POM3/control and control/POM3) were pooled.
Arm/Group | POM3 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 2/23 | 7/23
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | POM3 (N=23) | Placebo (N=23)
Allergy aggravated (General disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux (Gastrointestinal disorders) | 0 | 1
SGOT Increased (Hepatobiliary disorders) | 0 | 1
SGPT Increased (Hepatobiliary disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Purpura (Blood and lymphatic system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2
Decubitus Ulcer (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Ocular Hemorrhage (Eye disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Potential limitations: 1) relatively small sample size, and 2) relatively short length of wash-out period between treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No